CLINICAL TRIAL: NCT01973504
Title: A Multi-center, Multinational, Randomized, Double-blind, Controlled, Dose Comparison Study to Evaluate Safety and Efficacy of MP4OX Plus Standard Treatment, in Severely Injured Trauma Subjects With Lactic Acidosis Due to Hemorrhagic Shock
Brief Title: Phase 2c Dose Comparison Study of MP4OX in Trauma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sangart ceased operations
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRA-207
Record Dates: First submitted 2013-08-20; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Trauma; Hemorrhagic Shock; Lactic Acidosis
Keywords: Trauma; Hemorrhagic shock; Hemorrhage; Lactic acidosis; Oxygen therapeutics; Oxygen carriers; Ischemic rescue therapy; Hemoglobin solutions; PEGylated hemoglobin
MeSH Terms: conditions — Wounds and Injuries; Shock, Hemorrhagic; Acidosis, Lactic; Hemorrhage | interventions — polynitroxylated pegylated hemoglobin; maleimide-polyethylene glycol-modified hemoglobin, MP4; PEG-hemoglobin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MP4OX 500-mL (Experimental): 500-mL dose of MP4OX
  Interventions: Drug: MP4OX
- MP4OX 750-mL (Experimental): 750-mL dose of MP4OX
  Interventions: Drug: MP4OX
- Control (Sham Comparator): Standard crystalloid Keep Vein Open (KVO) infusion
  Interventions: Drug: Control

INTERVENTIONS:
Drug: MP4OX — 4.3 g/dL pegylated hemoglobin in balanced lactate-electrolyte solution
  Other Names: Hemoglobin pegylated; MalPEG-Hb; MP4; PEG-Hb; Pegylated-Hb
  Arms: MP4OX 500-mL; MP4OX 750-mL
Drug: Control — Crystalloid solution IV infusion drip to keep vein open
  Other Names: Keep vein open (KVO) infusion; Sham infusion
  Arms: Control

SUMMARY:
MP4OX is being developed as an ischemic rescue therapy to perfuse and oxygenate tissues at risk during hemorrhagic shock. MP4OX is a pegylated hemoglobin-based colloid designed to improve perfusion and target delivery of oxygen to ischemic tissues. This study will evaluate safety and efficacy of MP4OX treatment, in addition to standard therapy, in trauma patients suffering from lactic acidosis due to severe hemorrhagic shock.

DETAILED DESCRIPTION:
Acute trauma, including both blunt and penetrating injury, is often associated with uncontrolled bleeding that leads to hemorrhagic shock. During shock, inadequate blood flow results in local ischemia and tissue hypoxia (insufficient oxygenation) of critical organs with resulting lactic acidosis. More than 10% of trauma victims who reach hospital alive will die, and many will suffer from organ failure. The primary goal when treating traumatic hemorrhage is to control blood loss, support ventilation and oxygenation, and maintain cardiovascular function to maintain organ perfusion.

Despite optimal care, organ dysfunction is present in many patients as evidenced by persistent lactic acidosis. Blood transfusions are intended to improve circulation of oxygen-carrying red blood cells, but are frequently insufficient, even when the hemoglobin level is optimized. The severity of lactic acidosis in trauma victims has also been shown to correlate with worse outcome.

Support for the proposed application for MP4OX as a therapeutic adjunct to standard treatment of severe hemorrhage shock, is based on multiple preclinical studies in different animal models of hemorrhagic shock resuscitation. These preclinical studies demonstrated that survival was greater and restoration of acid-base status and hemodynamics were improved with MP4OX. The benefits of MP4OX in animals were observed with or without co-administration of autologous blood, demonstrating that red cell transfusion alone was insufficient, and that the effects of MP4OX were additive.

The hypothesis for the current study is that MP4OX will enhance perfusion and oxygenation of ischemic organs and thereby prevent and reduce the duration of organ failure and improve morbidity and mortality outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Trauma injury (blunt and/or penetrating) resulting in lactic acidosis due to hemorrhagic shock
* Acidosis (blood lactate level ≥ 5 mmol/L; equivalent to 45 mg/dL)

Exclusion Criteria:

* Massive injury incompatible with life
* Normalization of lactate prior to dosing (≤ 2.2 mmol/L)
* Evidence of severe traumatic brain injury (TBI) as defined by ANY one of the following: Known non-survivable head injury or open brain injury; Known AIS (head region) ≥ 4 by an appropriate imaging methodology; Contemplated CNS surgery; Abnormal physical exam indicative of severe CNS or any spinal cord injury above T5 level; or Glasgow Coma Score (GCS) = 3, 4 or 5.
* Cardiac arrest prior to randomization
* Known age below the legal age for consenting
* Estimated time from injury to randomization > 4 hours
* Estimated time from hospital admission to randomization > 2 hours
* Known pregnancy
* Use of any oxygen carrier other than RBCs
* Known previous participation in this study
* Professional or ancillary personnel involved with this study
* Known receipt of any investigational drug(s) within 30 days prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects discharged from hospital through Day 28 and alive at the Day 28 Follow up visit | 28 days

SECONDARY OUTCOMES:
Hospital-free, ICU-free, and Ventilator-free days | Through 28 and 60 days
Proportion of subjects remaining in hospital, ICU or on ventilator | Through 28 and 60 days
Days in hospital, in ICU, or on Ventilator | Through 28 and 60 days
All-cause Mortality | At 48 hours and 28 or 60 days
Time to discharge from ICU, hospital discharge, or liberation from ventilation | Through 28 or 60 days
Composite of Time to Complete Organ Failure Resolution (CTCOFR) | Day 21

OTHER OUTCOMES:
Daily modified Denver Score | Day 7
Proportion of patients with persistent renal dysfunction | Day 60
Duration of ICU stay for survivors | Day 28 and Day 60
Proportion of subjects who normalize lactate | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karim Brohi, MD, Principal Investigator — The Royal London Hospital; Frank V. Booth, BCh, FACS, Study Chair — Sangart, Inc.
Locations (31):
- Australia (2):
  - Liverpool Hospital, Liverpool
  - John Hunter Hospital, Newcastle
- Belgium (2):
  - Erasme University Hospital, Brussels
  - University Hospital Antwerpen, Edegem
- Brazil (3):
  - Faculdade de Medicina de S. J. Do Rio Preto, São José do Rio Preto
  - Hopital Universitário, Centro de Estudos em Emergências em Saúde, USP Ribeirão Preto, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo - FMUSP, São Paulo
- France (6):
  - Hôpital Beaujon, Clichy
  - Hôpital du Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Roger Salengro, CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Pitié-Salpêtrière, Paris
- Germany (5):
  - Universitätsklinikum der Rheinisch-Westfälische Technische Hochschule Aachen, Aachen
  - Campus Virchow Klinikum Charité Berlin, Berlin
  - Kliniken der Stadt Köln gGmbH Krankenhaus Merheim, Cologne
  - Klinikum der J.-W.-Goethe-Universität Frankfurt a.M., Franfurt
  - BG Klinik Ludwigshafen, Ludwigshafen
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Hadassah University Hospital, Ein-Karem, Jerusalem
- Auckland City Hospital, Auckland, New Zealand
- Oslo University Hospital Ullevaal, Oslo, Norway
- South Africa (5):
  - Netcare Union Hospital, Alberton
  - Vincent Palotti Dr Christiaan Barnard Memorial Hospital, Cape Town
  - Charlotte Maxeke Johannesburg Academic Hospita, Johannesburg
  - Netcare Milpark Hospital, Johannesburg
  - Chris Hani Baragwanath Hospital, Soweto
- Switzerland (2):
  - CHU Vaudois, Lausanne
  - UniversitätsSpital Zürich, Zurich
- The Royal London Hospital, London, United Kingdom

REFERENCES:
- [Background] Cole RH, Vandegriff KD. MP4, a vasodilatory PEGylated hemoglobin. Adv Exp Med Biol. 2011;701:85-90. doi: 10.1007/978-1-4419-7756-4_12. PMID 21445773
- [Background] Young MA, Lohman J, Malavalli A, Vandegriff KD, Winslow RM. Hemospan improves outcome in a model of perioperative hemodilution and blood loss in the rat: comparison with hydroxyethyl starch. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):339-47. doi: 10.1053/j.jvca.2008.08.006. Epub 2008 Oct 22. PMID 18948027
- [Background] Vandegriff KD, Winslow RM. Hemospan: design principles for a new class of oxygen therapeutic. Artif Organs. 2009 Feb;33(2):133-8. doi: 10.1111/j.1525-1594.2008.00697.x. PMID 19178457
- [Background] Vandegriff KD, Malavalli A, Mkrtchyan GM, Spann SN, Baker DA, Winslow RM. Sites of modification of hemospan, a poly(ethylene glycol)-modified human hemoglobin for use as an oxygen therapeutic. Bioconjug Chem. 2008 Nov 19;19(11):2163-70. doi: 10.1021/bc8002666. PMID 18837531
- [Background] Svergun DI, Ekstrom F, Vandegriff KD, Malavalli A, Baker DA, Nilsson C, Winslow RM. Solution structure of poly(ethylene) glycol-conjugated hemoglobin revealed by small-angle X-ray scattering: implications for a new oxygen therapeutic. Biophys J. 2008 Jan 1;94(1):173-81. doi: 10.1529/biophysj.107.114314. Epub 2007 Sep 7. PMID 17827244
- [Background] Cole RH, Vandegriff KD, Szeri AJ, Savas O, Baker DA, Winslow RM. A quantitative framework for the design of acellular hemoglobins as blood substitutes: implications of dynamic flow conditions. Biophys Chem. 2007 Jun;128(1):63-74. doi: 10.1016/j.bpc.2007.03.004. Epub 2007 Mar 13. PMID 17418478
- [Background] Young MA, Riddez L, Kjellstrom BT, Bursell J, Winslow F, Lohman J, Winslow RM. MalPEG-hemoglobin (MP4) improves hemodynamics, acid-base status, and survival after uncontrolled hemorrhage in anesthetized swine. Crit Care Med. 2005 Aug;33(8):1794-804. doi: 10.1097/01.ccm.0000172648.55309.13. PMID 16096458
- [Background] Drobin D, Kjellstrom BT, Malm E, Malavalli A, Lohman J, Vandegriff KD, Young MA, Winslow RM. Hemodynamic response and oxygen transport in pigs resuscitated with maleimide-polyethylene glycol-modified hemoglobin (MP4). J Appl Physiol (1985). 2004 May;96(5):1843-53. doi: 10.1152/japplphysiol.00530.2003. Epub 2004 Jan 16. PMID 14729723
- [Background] Winslow RM, Lohman J, Malavalli A, Vandegriff KD. Comparison of PEG-modified albumin and hemoglobin in extreme hemodilution in the rat. J Appl Physiol (1985). 2004 Oct;97(4):1527-34. doi: 10.1152/japplphysiol.00404.2004. Epub 2004 Jun 18. PMID 15208289
- [Background] Vandegriff KD, Bellelli A, Samaja M, Malavalli A, Brunori M, Winslow RM. Kinetics of NO and O2 binding to a maleimide poly(ethylene glycol)-conjugated human haemoglobin. Biochem J. 2004 Aug 15;382(Pt 1):183-9. doi: 10.1042/BJ20040156. PMID 15175010
- [Background] Tsai AG, Vandegriff KD, Intaglietta M, Winslow RM. Targeted O2 delivery by low-P50 hemoglobin: a new basis for O2 therapeutics. Am J Physiol Heart Circ Physiol. 2003 Oct;285(4):H1411-9. doi: 10.1152/ajpheart.00307.2003. Epub 2003 Jun 12. PMID 12805024
- [Background] Vandegriff KD, Malavalli A, Wooldridge J, Lohman J, Winslow RM. MP4, a new nonvasoactive PEG-Hb conjugate. Transfusion. 2003 Apr;43(4):509-16. doi: 10.1046/j.1537-2995.2003.00341.x. PMID 12662285
- [Background] McCarthy MR, Vandegriff KD, Winslow RM. The role of facilitated diffusion in oxygen transport by cell-free hemoglobins: implications for the design of hemoglobin-based oxygen carriers. Biophys Chem. 2001 Aug 30;92(1-2):103-17. doi: 10.1016/s0301-4622(01)00194-6. PMID 11527583
- [Background] Young MA, Riddez L, Kjellstrom BT, Winslow RM. Effect of maleimide-polyethylene glycol hemoglobin (MP4) on hemodynamics and acid-base status after uncontrolled hemorrhage in anesthetized swine: comparison with crystalloid and blood. J Trauma. 2007 Dec;63(6):1234-44. doi: 10.1097/TA.0b013e31815bd7b0. PMID 18212644
- [Background] Wettstein R, Tsai AG, Erni D, Winslow RM, Intaglietta M. Resuscitation with polyethylene glycol-modified human hemoglobin improves microcirculatory blood flow and tissue oxygenation after hemorrhagic shock in awake hamsters. Crit Care Med. 2003 Jun;31(6):1824-30. doi: 10.1097/01.CCM.0000069340.16319.F2. PMID 12794426
- [Background] Husain FA, Martin MJ, Mullenix PS, Steele SR, Elliott DC. Serum lactate and base deficit as predictors of mortality and morbidity. Am J Surg. 2003 May;185(5):485-91. doi: 10.1016/s0002-9610(03)00044-8. PMID 12727572
- [Background] Regnier MA, Raux M, Le Manach Y, Asencio Y, Gaillard J, Devilliers C, Langeron O, Riou B. Prognostic significance of blood lactate and lactate clearance in trauma patients. Anesthesiology. 2012 Dec;117(6):1276-88. doi: 10.1097/ALN.0b013e318273349d. PMID 23168430
- [Background] McNelis J, Marini CP, Jurkiewicz A, Szomstein S, Simms HH, Ritter G, Nathan IM. Prolonged lactate clearance is associated with increased mortality in the surgical intensive care unit. Am J Surg. 2001 Nov;182(5):481-5. doi: 10.1016/s0002-9610(01)00755-3. PMID 11754855
- [Background] Abramson D, Scalea TM, Hitchcock R, Trooskin SZ, Henry SM, Greenspan J. Lactate clearance and survival following injury. J Trauma. 1993 Oct;35(4):584-8; discussion 588-9. doi: 10.1097/00005373-199310000-00014. PMID 8411283
- [Background] Tsai AG, Cabrales P, Manjula BN, Acharya SA, Winslow RM, Intaglietta M. Dissociation of local nitric oxide concentration and vasoconstriction in the presence of cell-free hemoglobin oxygen carriers. Blood. 2006 Nov 15;108(10):3603-10. doi: 10.1182/blood-2006-02-005272. Epub 2006 Jul 20. PMID 16857991
- See also: Sangart Inc. (San Diego, CA) web site [Study SPONSOR] — http://www.sangart.com